CLINICAL TRIAL: NCT03831412
Title: CBT-I Versus ERRT: Impact on Sleep, Nightmares, and Suicidal Ideation
Brief Title: Cognitive Behavioral Therapy for Insomnia vs. Exposure, Relaxation, and Rescripting Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tulsa (Other)
Responsible Party: Principal Investigator, Joanne Davis, Professor, University of Tulsa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TU1802
Record Dates: First submitted 2018-10-27; First posted 2019-02-05 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Insomnia; Nightmare; Trauma
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Wounds and Injuries | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Active Comparator): 5 sessions of treating insomnia
  Interventions: Behavioral: CBT-I
- ERRT (Active Comparator): 5 sessions of treating post-trauma nightmares
  Interventions: Behavioral: ERRT

INTERVENTIONS:
Behavioral: CBT-I — Targeting insomnia symptoms to reduce suicidal ideation and sleep problems related to traumatic experience.
  Other Names: Cognitive Behavioral Therapy for Insomnia
  Arms: CBT-I
Behavioral: ERRT — Targeting post-trauma nightmares to reduce suicidal ideation and sleep problems related to traumatic experience.
  Other Names: Exposure, Relaxation, Rescripting Therapy
  Arms: ERRT

SUMMARY:
The objective of this project is to determine if directly addressing disturbed sleep and nightmares will impact client reports of suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* experiences at least one nightmare per week for the past month
* having previously experienced a traumatic event
* difficulty falling or staying asleep
* suicidal ideation
* actively under the care of another health care provider

Exclusion Criteria:

* untreated obstructive sleep apnea
* acute or apparent psychosis
* untreated or unstable bipolar disorder
* past history of seizure disorder or neurological disorder
* intellectual disability
* current substance dependence or in past 6 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | From initial assessment to each session of treatment, and at 3 and 6 months after treatment completion
  Change in frequency of insomnia symptoms
Change in Insomnia Severity Index | From initial assessment to each session of treatment, and at 3 and 6 months after treatment completion
  Change in severity of insomnia symptoms
Change in Sleep log | From initial assessment to each session of treatment, and at 3 and 6 months after treatment completion
  Change in frequency of nightmares
Change in Sleep log | From initial assessment to each session of treatment, and at 3 and 6 months after treatment completion
  Change in severity of nightmares
Change in Beck Suicide Scale | From initial assessment to each session of treatment, and at 3 and 6 months after treatment completion
  Change in severity of suicidal ideation

CONTACTS AND LOCATIONS:
Locations (1):
- Lorton Hall, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://nightmaretreatment.org